CLINICAL TRIAL: NCT00672529
Title: Orthomolecular Treatment as add-on Therapy for Childhood Asthma
Brief Title: Orthomolecular Therapy and Asthma in Children
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Canadian Institute of Natural and Integrative Medicine (Other)
Collaborators: Alberta Children's Hospital (Other); Alberta Health services (Other); Alberta Heritage Foundation for Medical Research (Other); SickKids Foundation (Other); Lotte & John Hecht Memorial Foundation (Other)
Responsible Party: Sabine Moritz, Director of Research, Canadian Institute of Natural and Integrative Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18376; NHPD 115797
Record Dates: First submitted 2008-05-05; First posted 2008-05-06 (Estimated); Last update posted 2011-02-04 (Estimated); Status verified 2011-02

CONDITIONS: Asthma
Keywords: Childhood Asthma; Inhaled Corticosteroids; Alternative Medicine; Vitamins, minerals, and fish oil as Add-on Treatment
MeSH Terms: conditions — Asthma | interventions — Orthomolecular Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Active Comparator)
  Interventions: Dietary Supplement: Orthomolecular Therapy or Placebo Comparator
- Placebo Group (Placebo Comparator)
  Interventions: Dietary Supplement: Orthomolecular Therapy or Placebo Comparator

INTERVENTIONS:
Dietary Supplement: Orthomolecular Therapy or Placebo Comparator — The custom formulation proposed in this study comprises Vitamins C, E, B6 and B12, magnesium, selenium, quercetin and fish oil in relatively large doses. It is not at present registered as a natural health product or drug product.
  Eligible patients will be randomized to an orthomolecular treatment regime or placebo with a 2:1 randomization ratio and will remain on their randomized treatment for 16 weeks. For the first 8 weeks of the intervention period inhaled corticosteroid treatment will be unchanged. In the remaining 8 weeks dose adjustment will occur every two weeks. Participants will be monitored closely for changes in their lung function.
  Other Names: CIN-AST-01

SUMMARY:
The purpose of this study is

1. To pilot the research methodology for a randomized trial on an orthomolecular treatment regime versus placebo as add-on therapy for children with asthma;
2. To obtain a preliminary estimate of the effectiveness of an orthomolecular treatment regime for allowing tapering of inhaled corticosteroids in clinically stable asthmatic children. The obtained estimate will allow sample size calculations for a full-scale randomized trial; and
3. To obtain preliminary information about the safety and tolerability of an orthomolecular treatment regime.

DETAILED DESCRIPTION:
An orthomolecular treatment approach that combines supplements has, to date, not been tested, although it is commonly used by naturopathic practitioners to treat respiratory problems in individual children. A well-designed controlled trial is needed to determine if this approach is effective. This smaller study should establish guidelines for a large trial to follow. This proposed research is particularly important, as the trend to use natural treatments may encourage non-compliance with conventional medical treatments, leading to poor asthma control.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 7 to 18 years
* Mild to moderate asthma diagnosed by a respirologist
* Use of budesonide at a dose of 200-800 µg/d (or equivalent corticosteroid therapy) for ≥3 months
* Stable asthma, defined as no significant change in the regular asthma medication and no acute asthma exacerbation requiring corticosteroid rescue for at least 3 months before enrollment in the run-in phase. Asthma symptoms must be under good control
* Baseline forced expiratory volume at 1 second (FEV-1) >= 70% of the predicted normal value.
* Possible participants treated with orthomolecular therapies within the previous year will require a wash out period of 7 days prior to enrolment in the trial. (Vitamin C > 200mg, Vitamin E >50IU, Vitamin B12 > 100µg, Magnesium > 200mg, Selenium > 50µg, Omega-3 > 300mg, Quercetin > 3mg, Vitamin B6 > 75mg will all be considered orthomolecular doses).

Exclusion Criteria:

* Known hypersensitivity to any component of the orthomolecular therapy or placebo.
* Acute infectious sinusitis or respiratory tract infection or active lung disease other than allergic asthma within 1 month or any other significant systemic disease within 3 months of the study entry visit.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
The last tolerated dose of inhaled corticosteroids will be the primary end point. | To safeguard against the possibility of excessive adverse events related to the tapering procedures or the orthomolecular treatment, an interim analysis will be conducted after 50% accrual is reached in this pilot investigation.

SECONDARY OUTCOMES:
The number (percentage) of patients with failed tapering and failed rescue will serve as secondary endpoint. | See primary endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Moritz, MSc, Principal Investigator — Canadian Institute of Natural and Integrative Medicine; Badri Rickhi, MB,BS,FRCPC, Principal Investigator — Canadian Institute of Natural and Integrative Medicine; Hude Quan, MD, PhD, Principal Investigator — University of Calgary; Sheldon Spier, MD,CM,FRCPC, Principal Investigator — Alberta Children's Hospital; Mary Noseworthy, MD, FRCPC, Principal Investigator — Alberta Children's Hospital; Eric Arrata, ND, Principal Investigator — Paradigm Health Group; Trevor Hoffman, ND, Principal Investigator — Paradigm Health Group; Paul Saunders, PhD, ND, Principal Investigator — Canadian College of Naturopathic Medicine; Sunita Vohra, MD,FRCPC,MSc, Principal Investigator — University of Alberta
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

REFERENCES:
- See also: Canadian Institute of Natural and Integrative Medicine, Calgary — http://www.cinim.org/